CLINICAL TRIAL: NCT01693224
Title: Feasibility of Using the Inverness Lateral Flow Urine LAM Test for Diagnosis of Tuberculosis in HIV-Positive TB Suspects in Cape Town, South Africa
Brief Title: Feasibility of a Lateral Flow Urine LAM Test for Diagnosis of Tuberculosis in South Africa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tuberculosis Clinical Diagnostics Research Consortium (Network)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMID 10-0051; NA_00043138 (Other: Johns Hopkins Medicine Institutional Review Boards)
Record Dates: First submitted 2012-09-23; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Miliary
Keywords: Tests, Diagnostic; Mycobacterium tuberculosis; Mycobacterium tuberculosis antigens; TB; Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Miliary; Lipoarabinomannan
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Miliary; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Alere "Determine" lateral-flow urine lipoarabinomannan assay — lateral-flow (point-of-care) urine test to detect the lipoarabinomannan (LAM) component of the M. tuberculosis antigen in the urine of TB suspects, in vitro.
  Manufacturer: Alere
  Other Names: Determine lateral-flow urine LAM TB test
Device: Alere "Clearview" ELISA urine LAM assay — ELISA-based urine test to detect the lipoarabinomannan component of the M. tuberculosis antigen in the urine of TB suspects, in vitro.
  Manufacturer: Alere.
  Other Names: Clearview ELISA urine LAM TB test
Device: Cepheid Xpert MTB/Rif assay
  Other Names: Cepheid Xpert MTB/Rif test

SUMMARY:
The purpose of this study is to evaluate the accuracy, diagnostic yield, operational performance, and time to diagnosis of a novel lateral-flow urine LAM test in detecting tuberculosis in HIV-infected adults.

A secondary study objective is to evaluate the accuracy and diagnostic yield of the Cepheid Xpert MTB/Rif test in detecting tuberculosis in the blood of HIV-infected adults.

DETAILED DESCRIPTION:
Background: Tuberculosis (TB) incidence and mortality have increased dramatically as a result of the HIV epidemic. In parts of sub-Saharan Africa, TB is the leading cause of death among HIV-infected patients and approximately 50% of TB patients are HIV co-infected. Early treatment of TB is hindered by the lack of rapid, accurate diagnostic modalities that can be applied in resource-constrained settings. Mycobacterial culture is the laboratory standard for diagnosis of active TB, but it is costly, requires access to specialized laboratories, and takes weeks to provide results. Sputum smear microscopy detects less than half of HIV-infected TB cases in many settings. The Global Plan to Stop TB has prioritized the development of simple, accurate, inexpensive tests for TB case detection in HIV-positive individuals.

LAM: As a strategy for rapid TB diagnosis, the detection of Mycobacterium tuberculosis antigens has been explored over several decades. Lipoarabinomannan (LAM), a glycolipid component of the outer cell wall of mycobacteria, is an attractive diagnostic target for several reasons: it is heat-stable; cleared by the kidney; detectable in urine; and as a bacterial product, has the theoretical potential to discriminate active TB from latent TB infection independent of human immune responses. A urine test could facilitate TB diagnosis in patients in whom sputum is uninformative or not obtainable, and lacks the infection-control risks associated with sputum production or blood collection. Urine LAM detection may be amenable to simple, rapid, inexpensive point-of-care platforms.

This is a prospective study to evaluate the accuracy, diagnostic yield, operational performance, and time to diagnosis of a novel lateral-flow urine LAM test in detecting tuberculosis in HIV-infected adults. HIV-positive adults suspected to have TB will be enrolled after providing informed consent. Urine will be obtained for testing using the novel lateral flow urine LAM assay and an existing ELISA-based urine LAM assay. Conventional microbiological tests for TB and chest x-rays will also be performed. These tests will be performed on all participants enrolled (target sample size = 500).

A secondary study objective is to determine the accuracy and diagnostic yield of the Cepheid Xpert MTB/Rif test in detecting tuberculosis in the blood of HIV-infected adults (the same set of participants on whom the LAM testing is done; approximate sample size = 500).

ELIGIBILITY:
Inclusion Criteria (Individuals must meet all of the following inclusion criteria in order to be eligible to participate):

* Informed consent
* Suspected active tuberculosis
* Willingness and ability to comply with study procedures
* Any one or more of the following:

  * Current cough
  * Fever at any time within the preceding 4 weeks
  * Night sweats at any time within the preceding 4 weeks
  * Weight loss within the preceding 4 weeks
* HIV-positive based on any one or more of the following:

  * written results of a positive HIV antibody test, and/or
  * written results of a positive HIV viral load, and/or
  * documentation in the medical record of positive HIV status by a treating clinician.

Exclusion Criteria (Any subjects meeting any of the following exclusion criteria at baseline will be excluded from study participation):

* Multidrug tuberculosis treatment for greater than two days within the previous 60 days
* Unwillingness or inability to provide a urine sample
* Known chronic pulmonary condition, e.g. asthma, chronic obstructive pulmonary disease, emphysema
* Respiratory distress, defined as respiratory rate of >30 or oxygen saturation <90%
* Any specific condition that in the judgment of the investigator precludes participation because it could affect a subject's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the lateral-flow urine LAM assay (LF-LAM) | One year
  * Conventional TB tests (mycobacterial blood & sputum culture) will be the reference standard used to calculate sensitivity of the LF-LAM test
  * Sensitivity is defined as TP/(TP+FN), or the number of true positives over (the number of true positives + the number of false negatives)
  * "true positive" = a positive LF-LAM result in a patient also having ≥1 culture positive for M. tuberculosis
  * "false negative" = a negative LF-LAM result in a patient also having ≥1 culture positive for M. tuberculosis
Failure rate of the lateral-flow urine LAM assay | One year
  Failure rate expressed as the proportion of lateral flow urine LAM tests that require repeating due to an unevaluable initial result
Inter-reader variability of the lateral-flow urine LAM assay | One year
  Expressed as the percent agreement
Specificity of the lateral-flow urine LAM assay (LF-LAM) | One year
  * Conventional TB tests (blood & sputum culture) will be the reference standard used to calculate specificity (Sp) of the LF-LAM
  * Sp=TN/(TN+FP), or #true negatives / (#true negatives + #false positives)
  * "true negative" = negative LF-LAM in "Not TB" patient
  * "false positive" = positive LF-LAM in "Not TB" patient
  * "Not TB" = meets all criteria below
    * no sputum/blood culture positive for MTB
    * no smear microscopy positive for acid-fast bacilli
    * no granulomas/caseous necrosis on histopathology
    * no clinical response to TB treatment
    * a plausible alternative diagnosis

SECONDARY OUTCOMES:
Sensitivity of the ELISA-based urine LAM test | One year
  * Conventional TB tests (mycobacterial blood & sputum culture) will be the reference standard used to calculate sensitivity of the ELISA LAM test
  * Sensitivity is defined as TP/(TP+FN), or the number of true positives over (the number of true positives + the number of false negatives)
  * "true positive" = a positive ELISA LAM result in a patient also having ≥1 culture positive for M. tuberculosis
  * "false negative" = a negative ELISA LAM result in a patient also having ≥1 culture positive for M. tuberculosis
Diagnostic yield (expressed as number of TB cases detected) of various diagnostic strategies (see description) | One year
  Diagnostic yield will be measured for strategies including a) lateral flow urine LAM testing plus sputum smear microscopy; b) ELISA urine LAM testing plus sputum smear microscopy; c) sputum smear microscopy plus sputum culture; d) sputum culture plus mycobacterial blood culture.
Time to diagnosis (expressed in days) of various diagnostic strategies (see description) | One year
  Time to diagnosis will be measured for strategies including a) lateral flow urine LAM testing plus sputum smear microscopy; b) ELISA urine LAM testing plus sputum smear microscopy; c) sputum smear microscopy plus sputum culture; d) sputum culture plus mycobacterial blood culture.
Accuracy, efficiency, costs, and cost-effectiveness of various combinations of TB diagnostic tests | One year
  TB diagnostic tests to be included in this analysis: sputum smear microscopy, sputum culture, mycobacterial blood culture, chest X-ray, lateral-flow urine LAM testing, ELISA urine LAM testing, and Xpert MTB/Rif.
Satisfaction of lateral-flow urine LAM test operators | One year
  Based on questionnaire assessment
Specificity (Sp) of the ELISA-based urine LAM test | One year
  * Conventional TB tests (blood & sputum culture) will be the reference standard used to calculate Sp of ELISA LAM
  * Sp=TN/(TN+FP), or #true negatives / (#true negatives + #false positives)
  * "true negative" = negative ELISA LAM in "Not TB" patient
  * "false positive" = positive ELISA LAM in "Not TB" patient
  * "Not TB" = meets all criteria below
    * no sputum/blood culture positive for MTB
    * no smear microscopy positive for acid-fast bacilli
    * no granulomas/caseous necrosis on histopathology
    * no clinical response to TB treatment
    * a plausible alternative diagnosis
Sensitivity of the Xpert MTB/Rif test to detect MTB in blood | One year
  Conventional mycobacterial blood culture will be the reference standard used to calculate sensitivity of Xpert MTB/Rif in blood
  * Sensitivity is defined as TP/(TP+FN), or the number of true positives over (the number of true positives + the number of false negatives)
  * "true positive" = a positive Xpert MTB/Rif result in a patient also having ≥1 mycobacterial blood culture positive for M. tuberculosis
  * "false negative" = a negative Xpert MTB/Rif result in a patient also having ≥1 mycobacterial blood culture positive for M. tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dorman, MD, Study Chair — Johns Hopkins University; Mark Nicol, MBChB, PhD, Principal Investigator — University of Cape Town, Faculty of Health Sciences, Dept. of Medical Microbiology, Cape Town, South Africa; Mischka Moodley, MBChB, DTM&H, FCPath(Micro)SA, Principal Investigator — University of Cape Town, Faculty of Health Sciences, Dept. of Medical Microbiology, Cape Town, South Africa
Locations (2):
- South Africa (2):
  - G.F. Jooste Hospital, Cape Town, Western Cape
  - Town Two Clinic, Cape Town, Western Cape

REFERENCES:
- [Derived] Nakiyingi L, Moodley VM, Manabe YC, Nicol MP, Holshouser M, Armstrong DT, Zemanay W, Sikhondze W, Mbabazi O, Nonyane BA, Shah M, Joloba ML, Alland D, Ellner JJ, Dorman SE. Diagnostic accuracy of a rapid urine lipoarabinomannan test for tuberculosis in HIV-infected adults. J Acquir Immune Defic Syndr. 2014 Jul 1;66(3):270-9. doi: 10.1097/QAI.0000000000000151. PMID 24675585